CLINICAL TRIAL: NCT01005589
Title: Measurement of Neutrophil Membrane CD64 as an Early Indication of Neonatal Infection and Necrotising Enterocolitis (NEC).
Brief Title: CD64 Measurement in Neonatal Infection and Necrotising Enterocolitis
Status: Completed | Type: Observational
Sponsor: Newcastle-upon-Tyne Hospitals NHS Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 5026; 09/H0905/58
Record Dates: First submitted 2009-10-30; First posted 2009-11-02 (Estimated); Last update posted 2017-04-07 (Actual); Status verified 2017-04

CONDITIONS: Neonatal SEPSIS; Enterocolitis, Necrotizing
Keywords: Neonatal sepsis; Necrotizing enterocolitis; CD64 antigen; Receptors, IgG
MeSH Terms: conditions — Neonatal Sepsis; Enterocolitis, Necrotizing

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Bacterial infections are a major cause of death in newborn infants. And are linked to complications including: sepsis (an over exaggerated immune response to infection) and necrotising enterocolitis (a potentially fatal inflammatory bowel disease).

Detecting infections at an early stage is difficult in newborns as the signs and symptoms can be non-specific, the most commonly used lab test is to culture a sample of blood, urine or spinal fluid to try and grow and identify any bacteria that is present; however these tests take 24-48 hours to give results, and this means that neonates who present with signs of infection are prescribed broad spectrum antibiotics whilst results are obtained.

The lack of a test that can detect infection at an early stage and give rapid results is one of the major problems in the diagnosis and management of infection in newborns. This study will investigate neutrophils, which are white blood cells that are important in fighting infection. When neutrophils detect and infection they become activated, and produce a protein called CD64 (a cell marker) on their surface, and it is this protein that we want to measure. Neutrophils produce the CD64 protein within 1 hour of first detecting an infection, so we could hopefully detect and treat infections much quicker.

The hypothesis this study will test are:

1. Does neutrophil membrane CD64 measurement provide a highly sensitive and specific marker of infection in neonates AND:
2. Does neutrophil membrane CD64 measurement provide a highly sensitive and specific marker of NEC in neonates

DETAILED DESCRIPTION:
New born infants (neonates) and particularly premature infants are more at risk of developing bacterial infections due to a number of different factors including immature immune systems, and because they are more likely to need invasive procedures such as chest drains that increase the potential for infection.

The signs of infection in babies can be non-specific and difficult to diagnose. Undetected infections which are not treated can quickly lead to sepsis, which is an over-exaggerated response by the immune system which can spread throughout the whole body and attack 'self' tissue leading to organ failure and death. It is therefore vital that infection in neonates can be diagnosed quickly in order to administer the best treatment.

The current 'gold standard' laboratory test for detecting infection is to culture samples of blood, urine or spinal fluid, which allows any bacteria present to be grown in the lab and identified. However this test can take 24-48 hours to give results, and due to the devastating consequences of not treating an infection in neonates it is now common practice to prescribe broad spectrum antibiotics to any neonate who presents with signs of infection and await test results.

This study will look at what happens to the white blood cells that make up part of the immune defence against infection when they encounter an infection. One type of white blood cell that is particularly important in fighting bacterial infections is called the neutrophil, and when it detects an infection, it becomes activated in order to fight it; during this activation process it expresses a protein marker called CD64 on its surface. The CD64 protein is expressed within hours of the onset of bacterial infections, so measuring the CD64 marker could provide much faster results than laboratory tests that are currently available.

If we could detect infections in neonates more rapidly then non-infected neonates (with negative CD64 result) could have antibiotic treatment stopped. This is beneficial as it reduces unnecessary treatment therefore reducing hospital stays and cost. It also reduces the use of antibiotics, the overuse of which can promote the development of antibiotic resistant strains of bacteria, which can colonize entire wards. It would also mean that infected neonates could receive more appropriate care, for example more specific antibiotics.

Necrotising enterocolitis (NEC) is another common condition that affects newborn infants. Exactly how and why some infants develop NEC is still unclear, but is thought to be due to a number of different factors including bacterial infection. Advanced NEC is characterised by bowel necrosis, bowel perforation, sepsis and death and remains one of the major causes of morbidity and death in neonates, with a mortality rate of 30-50%.

The diagnosis of NEC is currently based on X-ray findings and features such as air in the abdomen are very diagnostic. Other biochemical and haematological parameters are also used to support X-ray findings. Because we know that one of the 'triggers' for the initiation of the disease is a bacterial infection: culturing samples of blood, urine or spinal fluid is important to try and identify/isolate any infection. However these tests all take time, and current practice means that any neonate who presents with signs of NEC/infection will be subjected to gut rest i.e. nil by mouth (in order to prevent any further damage to the gut) and also be prescribed broad spectrum antibiotics. Patients who have suspected NEC will often be continued on a treatment/monitoring regime, the length of which will be dictated by clinical judgment: and this may be unnecessary if there is no sign of infection/inflammation.

One of the greatest challenges in the management/diagnosis of NEC is the lack of an early, reliable and consistent marker of 'intestinal inflammation' in peripheral blood. This study will investigate if the CD64 marker can fill this gap.

The inflammatory process seen in NEC is probably initiated by the presence of bacteria. The bacteria activate cells of the innate immune system which produce a number of inflammatory mediators causing inflammation. The CD64 marker is not a 'direct' marker of inflammation, however the cells that are activated in order to produce inflammation i.e. neutrophils will be positive for CD64 once activated, therefore if CD64 is not present on the cells: they have not been activated, which means there is no infection and therefore no inflammation.

If the CD64 marker can rule out infection in neonates with suspected NEC, then it also rules out any ongoing inflammatory process. Clinicians could use the CD64 assay in conjunction with X-ray findings in order to stop treatment in non affected neonates and restart feeding sooner, which has many benefits to the neonate's growth and nutritional development, and also negates the need for prolonged antibiotic treatment and hospital stays. It also means that affected neonates could receive more appropriate treatment and monitoring.

Taking serial (repeated) measurements from patients with suspected or confirmed NEC at various intervals (24 48 hours etc.) and seeing how this compares with the clinical picture, could possibly be used to monitor the disease progression/severity e.g. could a rapid rise in the expression of CD64 indicate progression to the advanced stage and need for surgery, and could a reduced expression of CD64 indicate remission or response to treatment.

ELIGIBILITY:
Inclusion Criteria:

* Clinical suspicion of infection / NEC
* In patient on ward 35 at RVI (neonatal ward)
* Male or Female
* Parental consent obtained
* Neonate

Exclusion Criteria:

* Known congenital abnormalities (Downs syndrome, leukaemia)
* Parental consent not obtained

Max Age: 1 Month | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Patients from the neonatal ward who have suspected infection/NEC will be recruited into the study.
Sampling Method: Non-Probability Sample
Enrollment: 59 (Actual)
Dates: Start 2009-10; Primary Completion 2010-06-02 (Actual); Study Completion 2010-06-02 (Actual)

PRIMARY OUTCOMES:
The primary outcome measure is the CD64 count at the time of presentation with symptoms of infection/NEC. | At time of initial sepsis evaluation

CONTACTS AND LOCATIONS:
Overall Officials: Janet E Berrington, Principal Investigator — Newcastle upon Tyne NHS Foundation Trust
Locations (1):
- Newcastle upon Tyne NHS foundation Trust, Newcastle, Newcastle-upon-Tyne, United Kingdom